CLINICAL TRIAL: NCT02575742
Title: Colonic Motility And Gut Microbiota Composition In Constipation And Ageing
Brief Title: Colonic Motility in Constipation and Ageing
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: ReDA-010366 QM
Record Dates: First submitted 2015-09-15; First posted 2015-10-15 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2015-10

CONDITIONS: Ageing; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Young women without chronic constipation: Healthy women without chronic constipation who are aged between 18-40 years
  Interventions: Device: 3D-Transit system
- Older women without chronic constipation: Healthy women without chronic constipation who are aged between 70-90 years
  Interventions: Device: 3D-Transit system
- Young women with chronic constipation: Women with symptoms of chronic constipation who are aged between 18-40 years
  Interventions: Device: 3D-Transit system
- Older women with chronic constipation: Women with symptoms of chronic constipation who are aged between 70-90 years
  Interventions: Device: 3D-Transit system

INTERVENTIONS:
Device: 3D-Transit system

SUMMARY:
The reason chronic constipation (CC) becomes commoner with age is not fully understood. New studies suggest that bowel contraction patterns, dietary fibre and gut bacteria are important and may differ in older people. Since CC reduces quality of life and is a major reason why elderly are admitted to hospitals and residential care, there is a need to understand how these factors change with age.

Currently, placing a pressure sensing catheter inside the large intestine (pancolonic manometry) is the gold standard way to measure how well it contracts. However this involves a camera test (colonoscopy) which is invasive with risks of bowel perforations (~80/100,000). The risk is higher with age (64-80yr: ~90/100,000; 80+yrs: ~120/100,000), making it unethical for elderly.

A technique called the 3D-Transit System has been developed, involving a small ingestible capsule, containing a 'trackable' electromagnet. By tracking movements of the capsule swallowed by participants, it provides precise detailed information on the capsule progression inside the whole gut and large bowel's contractile activity in real-time. It is minimally-invasive and radiation-free, making it possible to assess elderly for the first time.

This study aims to assess how bowel contraction patterns, dietary fibre intake and gut bacteria differ between young and older adults (with and without CC), to better understand why CC is more common in elderly.

It is a pilot, 4 arm, single centre, observational study involving 60 women aged 18-40 years and 70-90 years (15 non-constipated and 15 with CC for each age group). The study lasts 3 weeks, containing 2 weeks of run-in period and 1 week of study period.

The four groups participants will be asked to: swallow 2 capsules to assess their large bowel's contractile function using the 3D-transit system; provide stool samples to analyses their gut bacteria; and complete questionnaires to assess their gastrointestinal symptoms.

DETAILED DESCRIPTION:
Type of study Experimental study comparing colonic contractile functions (including region-specific gut transit times) between healthy young vs. older women, and between constipated young women vs. constipated older women

Design 4-arm observational pilot study

Study Population The study will include 15 healthy young women, 15 healthy older women, 15 young women with chronic constipation and 15 older women with chronic constipation (but otherwise healthy). Vulnerable subject groups (e.g. elderly with dementia) will not be included.

Subject Recruitment Participants with constipation will be identified mainly from the existing database of patients with constipation who had previously participated in research or undertaken anorectal physiology investigations at the GI physiology unit (part of Queen Mary University of London). [The GI physiology unit is part of an academic institution (Queen Mary University of London) and not part of the NHS. However being a specialised centre for anorectal physiological assessments, it investigates patients referred from various NHS sites throughout the UK. Thus it has built up a database of individuals with constipation who had previously undergone anorectal examinations and/or research]. Suitable participants will be identified by the Director (also Chief Investigator for this study) and staff of the GI physiology unit, who have access to the database and patients' medical records and personal data. Following identification, an invitation letter (containing the research team's contact details) will be sent to patients by the director of the unit (see supporting document). Potential participants with constipation will also be recruited via advertisement.

Participants without constipation will be recruited using mailing lists of public involvement groups. Participants will also be recruited through advertisements, posters, and/or websites in local media, social media, websites, academic institution, medical institutions and GP surgeries. The same text and layout will be used for all forms of advertising.

Participants who contact us to express interest will be asked to provide us their contact details so that we can send them details of the study including the participant information sheet.

Participants will be asked to read this information sheet and to contact us if they require any clarification or further explanations. Participant will be asked to take as long as they wish to consider the information given and if they wish, to discuss with any family, friends, GP or INVOLVE [(http://www.invo.org.uk/) a national advisory group that supports greater public involvement in NHS, public health and social care research, who share knowledge and learning on public involvement in research]

Participants who would like to participate after reading the study information sheet will be asked to contact us again to arrange a date for a pre-screening telephone call.

For participants who met the criteria during pre-screening, a date for the screening visit will be arranged where full screening will take place.

After the study is explained in detail to the subjects at the study site during the screening visit (V1, see below), and they have agreed to participate by signing the written informed consent form, an eligibility checklist will be completed.

Volunteers will be compensated for their participation in the study and travel expenses will be reimbursed.

Study visits Initial pre-screening (by telephone) On the agreed day, a qualified member of the research team will make a phone call to individuals who are interested in participating in the study after reading the participant information sheet. Verbal consent will be obtained and potential participants will be pre-screened against the main inclusion and exclusion criteria.

Screening V1 (study day -14)

At V1, a full screening will be performed in person to evaluate eligibility according to the criteria. Assessments will include evaluation of:

* Medical and surgical history
* Symptoms of constipation, using a screening questionnaire detailing American College of Gastroenterology definition of constipation, the CCCS questionnaire and Bristol Stool Scale. (Subjects will be asked to complete other questionnaires such as PAC-SYM and HADS at the baseline visit - see below).
* Concomitant diseases
* Current medications, particularly treatments used for symptoms of constipation within the past 12 weeks
* Barthel index (See supporting document)
* Pregnancy status of the women subjects with child-bearing potential, using urinary pregnancy tests. Appropriate advice will be given to all women of potential child-bearing age stating that they must be willing to use a 'highly effective' method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until completion of the study.
* Abdominal diameter, measured as the circumference at the level of the umbilicus

For eligible subjects:

* Written informed consent & participant demographic data will be obtained
* Subjects will be instructed to start a 2 week run in period, during which they will continue with their usual diet, physical activity but will discontinue use of laxative, prokinetics, probiotics, prebiotics, or fibre supplements until the end of the study.
* Subjects will be instructed to read food labels carefully to check the content for addition of probiotics or prebiotics. Subjects are permitted to use Bisacodyl or glycerine suppositories as rescue laxatives if they had not had a bowel movement for 4 or more days and experienced abdominal discomfort; its use needs to be documented on the stool diaries.
* Baseline visit will be scheduled. To eliminate the potential effect of hormonal changes on bowel function, baseline date will be synchronized to the menstrual cycle for premenopausal women (subjects to start in the midfollicular phase [days 6 - 8 of the menstrual cycle].
* Subjects will be asked to collect a single fresh stool sample and bring it to the study centre either on the baseline visit day or anytime during the 5 days prior to the baseline visit, provided that the sample is transferred to the study centre within 3 hours of collection. Stool samples collected during the study will be initially handled at Queen Mary University of London. Samples will be sent from the chief investigator (Dr Mark Scott, Wingate Institute, 26 Ashfield Street, E1 2AJ, Queen Mary University of London) to King's College London (Professor Kevin Whelan, Diabetes and Nutritional Sciences Division, 150 Stamford Street, SE1 9NH), and Nestle Research Centre (Dr Peter Duncan, PO Box 44, CH-1000, Lausanne 26, Switzerland) for further stool microbiology analysis. All experimental material will be destroyed at the end of the study.
* Subjects will be asked to complete a daily bowel diary for 1 week and a food diary for 3 days (Sat, Mon, Tue) before baseline visit.

  * For elderly participants who have difficulties attending the study centre, study staff will perform the subsequent visits at the participants' home (following consent). This will be considered on an individual basis.

Baseline V2 (study day 0) On the day of the experiment (study day 0), participants will visit the study centre at 8 am after an overnight fast. The participants will be provided with a standardized breakfast snack and the detector will be attached. Capsules (capsule 1 and capsule 2) will be activated and communication between the capsules and the detector will be confirmed. Immediately afterwards, capsule 1 will be swallowed with a glass of water at 8 am. Subjects will then be asked to complete the following questionnaires before leaving the study centre: St Mark's Incontinence scale, PAC-QOL, PAC-SYM, SF12 and HADS. Questionnaire entries will be reviewed immediately by the investigator upon collection

Participants will also be asked to keep a second bowel diary and a record of their meal times during the study period.

The participants will be instructed not to eat again for six hours to avoid prolongation of gastric emptying. Throughout the study period, participants will be allowed to perform most of their normal daily activities, including taking public transportation and going to work. Hard physical activities (work and all sports) will be prohibited. They will also be asked to wear the detector vest at all times throughout the study. The detector vest will only be taken off for a few minutes each morning to allow participants to take a shower.

All potential adverse events / serious adverse events and changes in concomitant diseases / medications since the screening visit will be monitored throughout the study period.

Study period V3 (study day 1) After an overnight fast, participants will visit the study centre at 8 am. Participants will be provided with a standardized breakfast snack and asked to swallow the second capsule (capsule 2). The study staff will perform a review of any adverse events. The participants will be instructed not to eat again for six hours following ingestion of the capsule to avoid prolonging gastric emptying.

Study period V4 (any between Day 2 and Day 6):

Participants will be asked to return to the study centre when they have a bowel movement and observed that both capsules (1 & 2) have been expulsed from the body with their faeces. If participants have not defaecated after 5 days have elapsed following ingestion of the last capsule, they will be also asked to return to the study centre.

During this visit, the study staff will download the data from the detector vest and check if any of the capsules remain in the participants' gastrointestinal tract using a laptop and the software for the ambulatory 3D-transit system.

The study's end date is dependent on the retention time of both capsules. The study will terminate if:

1. It has been confirmed that both capsules have exited the body; or
2. 5 days have elapsed since ingestion of the last capsule (maximum battery life of each capsule is 5 days), whichever occurs earlier.

The detector will be removed when the study is terminated. In non-constipated subjects (who defaecate at least 3 times per week as defined by the inclusion / exclusion criteria), the study is anticipated to end 3 days after ingestion of the second capsule (at the latest). In constipated participants (who defaecate <3 times per week as defined as defined by the inclusion / exclusion criteria), the study is anticipated to end 5 days after ingestion of the second capsule (at the latest).

For subjects who still have one or both of the capsules remaining in the gastrointestinal tract during V4, the research team will perform telephone follow up to check if participants have developed any abdominal symptoms until the participants have a bowel opening and observe that both capsules (capsule 1 & 2) have been expulsed from the body.

Study duration The duration of the study for each subject will be 3 weeks. This is comprised of 2 weeks of run-in period (following screening & enrolment) and a maximum of 1 week of study period (following capsule ingestion).

ELIGIBILITY:
Inclusion criteria for constipated group

* Aged 18-40 or 70-90 years of age
* Barthel index ≥11 [for elderly women only]
* No co-existing acute or chronic diseases at the time of recruitment (except hypertension and hypercholesterolemia for elderly women)
* Patients with self-reported problematic constipation
* Cleveland Clinic Constipation Score ≥8
* Bowel movement frequency <3 per week
* Stool consistency of 1-3 on the Bristol Stool Chart
* No evidence of organic causes of constipation
* Symptoms of constipation (unsatisfactory defaecation characterized by infrequent stool, difficult stool passage or both for at least the previous 3 months)

Inclusion criteria for non-constipated group

* Healthy women aged 18-40 or 70-90 years of age
* No co-existing acute or chronic diseases at the time of recruitment (except hypertension and hypercholesterolemia for elderly women)
* Barthel index ≥11 [for elderly women only]
* Cleveland Clinic Constipation Score <8

Exclusion Criteria:

* Inability to understand written and spoken English
* Lacking capacity to understand subject information sheet and give informed consent
* Vulnerable subject groups (e.g. elderly with dementia)
* Pregnancy, intention to become pregnant, or breastfeeding during study period
* Recent childbirth in the last 6 months
* Other causes of reduced / dysregulated GI motility and secondary constipation
* Conditions which make it unsafe to use the capsules

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 women aged 18-40 years (15 non-constipated women, 15 with chronic constipation) and 30 women aged between 70-90 years (15 non-constipated women, 15 with chronic constipation) will be recruited, via advertisement in the community.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Total colonic transit time | 2 to 5 days
  Colonic transit time as measured by 3D transit system

CONTACTS AND LOCATIONS:
Overall Officials: Mark Scott, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom